CLINICAL TRIAL: NCT04087135
Title: Comparison of the Success Rate of Intubation With Direct Laryngoscopy or Videolaryngoscopy in an Hemoptysis Simulated Situation on Human Cadaver Embalmed With Thiel's Method
Brief Title: Comparison of Intubation With Direct Laryngoscopy or Videolaryngoscopy in an Hemoptysis Simulated Situation on Human Cadaver Embalmed With Thiel's Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Centre d'Apprentissage des Habiletés Cliniques (CAAHC) (Unknown); Laboratoire d'anatomie de Trois-Rivières (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: HP2018
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2018-10

CONDITIONS: Laryngoscope; Hemoptysis; Simulation; Cadaver; Intubation; Difficult or Failed
Keywords: videolaryngoscopy; Thiel's embalmed cadaver
MeSH Terms: conditions — Hemoptysis; Cadaver | interventions — Suction

STUDY DESIGN:
Intervention Model Description: Each participant will performe the intubation three time using the tools provided, for the same simulation situation: (a) direct laryngoscopy, (b) videolaryngoscopy McGrath and (c) videolaryngoscopy McGrath with suction.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- participant LD (Experimental)
  Interventions: Other: direct laryngoscopy
- participant VL (Experimental)
  Interventions: Other: videolaryngoscopy McGrath
- participant VLS (Experimental)
  Interventions: Other: videolaryngoscopy McGrath with suction

INTERVENTIONS:
Other: direct laryngoscopy — Participants will intubate the hemoptysis cadaver model in simulation with direct laryngoscopy MacIntosh blade.
  Arms: participant LD
Other: videolaryngoscopy McGrath — Participants will intubate the hemoptysis cadaver model in simulation with videolaryngoscopy using McGrath and the short curved blade (XBlade)
  Arms: participant VL
Other: videolaryngoscopy McGrath with suction — Participants will intubate the hemoptysis cadaver model in simulation with videolaryngoscopy using McGrath and the short curved blade (XBlade) and a suction they will advanced directly before the optic of the camera.
  Arms: participant VLS

SUMMARY:
Our study first aims to develope a realistic cadaver model of hemoptysis based on Thiel's embalmed cadavers. Secondly, participants will intubate the hemoptysis cadaver model with (a) the direct laryngoscopy with MacIntosh blade, (b) the videolaryngoscopy with McGrath XBlade and (c) the videolaryngoscopy with McGrath XBlade and a suction advance before the optic of the camera. We hypothesis that, in simulated hemoptysis on the Thiel's embalmed cadaver, the rate of failed intubation at first try will be different depending on the laryngoscope used.

DETAILED DESCRIPTION:
For the simulation of hemoptysis, we will need to use the Thiel's embalmed cadaver, who's realism is established, create a synthetic form of blood resembling real blood by its viscosity and color for the simulation and elaborate the dynamic interface of the simulation of hemoptysis. The quantity and way of administration of the blood through the trachea will be tested to obtain a realistic hemoptysis as seen in supraglottic.

For the simulation, we will compare the efficiency of intubation, judged by the failure rate of intubation on first try, for (a) the direct laryngoscopy with MacIntosh blade, (b) the videolaryngoscopy with McGrath XBlade and (c) the videolaryngoscopy with McGrath XBlade with the suction advanced before the camera. We will also measure the time to intubation, the failure rate of intubation, the suction use and the difficulty of intubation as reported by the participants.

ELIGIBILITY:
Inclusion Criteria:

* all wiling doctors and medical residents in the departments of anesthesiology, emergency medicine and intensive care
* experience with the technique of intubation using videolaryngoscopy and direct laryngoscopy.

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
failure of intubation on first try | the duration of the simulation
  defined as the withdrawal of the laryngoscope from the mouth

SECONDARY OUTCOMES:
time to intubation | the duration of the simulation
  from the insertion of the laryngoscope in the mouth to the inflation of the endotracheal cuff
failure in intubation | the duration of the simulation
  failure to intubate after three try
use of suction | the duration of the simulation
  document the use of suction
difficulty of intubation | the duration of the simulation
  as describe by the participants on a Likert scale 1 to 5

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided